CLINICAL TRIAL: NCT01346397
Title: Prospective Randomized Trial Comparing CsA Versus Tacro After Campath Induction In Kidney Transplant Recipients
Brief Title: Study Cyclosporine (CsA) Versus Tacrolimus (Tacro) After Campath Induction in Kidney Transplantation
Acronym: RSCS-Campath
Status: Completed | Type: Observational
Sponsor: Russian Academy of Medical Sciences (Other)
Collaborators: Russian Scientific Center of Surgery (Unknown)
Responsible Party: Principal Investigator, Michael Kaabak, professor, Russian Academy of Medical Sciences
Other Study IDs: RSCS-Campath-06
Record Dates: First submitted 2010-07-07; First posted 2011-05-03 (Estimated); Results first posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: Acute Graft Rejection; Chronic Allograft Nephropathy; Polyomavirus-related Transplant Nephropathy
Keywords: rejection; survival; alemtuzumab; cyclosporine; tacrolimus
MeSH Terms: conditions — Rejection, Psychology | interventions — Cyclosporine; Tacrolimus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — blood and urine, taken at the time of protocol or case biopsies will be deeply freeze and stocked for future examination for NAT or other molecules - candidates for diagnostic markers.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- cyclosporine group: cyclosporine group - after alemtuzumab induction cyclosporine was administered
  Interventions: Drug: cyclosporine or tacrolimus
- tacrolimus group: tacrolimus group - after alemtuzumab induction tacrolimus was administered
  Interventions: Drug: cyclosporine or tacrolimus

INTERVENTIONS:
Drug: cyclosporine or tacrolimus — after alemtuzumab, cyclosporine or tacrolimus was administered

SUMMARY:
After alemtuzumab induction, followed with kidney transplantation, patients will be randomly assigned to receive either tacrolimus or cyclosporine microemulsion in combination with mycophenolates. Patients will be followed including protocol biopsy at 1, 12, 36, 60 month posttransplant, regular nuclein acid testing (NAT) for cytomegalovirus (CMV), Epstein-Barr virus (EBV) and BK virus (BKV) in urine and blood.

The investigation is undertaken to clarify the reason for equal survival rates for patients on cyclosporine and tacrolimus despite the lower rejection rate on tacrolimus.

DETAILED DESCRIPTION:
Special attention will be paid to the epidemiology of virus infections behind one year post transplant. Very limited data are available on this issue and there is suspicion that tacrolimus patients suffer more hard with viruses like CMV, EBV, BKV. These viruses can induce graft nephropathy and threat to the life of the recipient.

ELIGIBILITY:
Inclusion Criteria:

* first kidney allograft recipients
* alemtuzumab induction

Exclusion Criteria:

* CNI intolerance

Ages: 6 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Recipients of kidney allograft who underwent previous Campath induction and do receive calcineurine inhibitor (CNI)
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2009-04; Primary Completion 2013-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Kaabak, professor, Principal Investigator — Russian Scientific Center of Surgery RAMS
Locations (1):
- National Research Centre of Surgery, Moscow, Russia

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyclosporine Group: cyclosporine group - after Campath induction cyclosporine will be administered
- Tacrolimus Group: tacrolimus group - after Campath induction tacrolimus will be administered
Period: Overall Study
Arm/Group | Cyclosporine Group | Tacrolimus Group
Started | 85 | 85
Completed | 85 | 85
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclosporine Group | Tacrolimus Group | Total
Number analyzed (Participants) | 85 | 85 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 19 (14) | 21 (15) | 20 (14)
Gender [Number; unit: participants]
  Female | 33 | 35 | 68
  Male | 52 | 40 | 92
Deceased donor kidney transplant recipients [Number; unit: participants] | 28 | 21 | 49

OUTCOME MEASURES:

1. Primary Outcome: Patient Survival
Description: in cyclosporine group 96.4 +/- 2.8%; in tacrolimus group 96.3 +/- 3.4%
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine Group | Tacrolimus Group
Number analyzed (Participants) | 85 | 85
percentage of participants | 96.4 [94 to 98.8] | 96.3 [92.9 to 99.7]

2. Primary Outcome: Graft Survival
Description: in cyclosporine group 84.6 +/- 5.8%; in tacrolimus group 86.2 +/- 4.1%
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine Group | Tacrolimus Group
Number analyzed (Participants) | 85 | 85
percentage of participants | 84.6 [78.7 to 90.5] | 86.2 [82.6 to 93.5]

ADVERSE EVENTS:
Arm/Group | Cyclosporine Group | Tacrolimus Group
Serious Adverse Events (participants affected / at risk) | 13/85 | 12/85
Other Adverse Events (participants affected / at risk) | 40/85 | 12/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclosporine Group (N=85) | Tacrolimus Group (N=85)
kidney graft loss (Renal and urinary disorders) | 9 (9) | 9 (9)
patient death (Cardiac disorders) | 4 (4) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclosporine Group (N=85) | Tacrolimus Group (N=85)
clinical acute rejection (Immune system disorders) | 30 (30) | 7 (7) — rejection accompanied by disturbances of the kidney graft function
all rejection rate, including subclinical rejections. (Renal and urinary disorders) | 40 (40) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes